CLINICAL TRIAL: NCT03027999
Title: Efficiency of a Tight Monitoring by a Nurse Practitioner of Rheumatoid Arthritis (RA) Patients in Remission (or Low Disease Activity) Under Rituximab to Detect Early Relapse of the Disease
Brief Title: Efficiency of a Tight Monitoring by a Nurse Practitioner of Rheumatoid Arthritis (RA) Patients in Remission
Acronym: SIERRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/0190/HP
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituximab; tight monitoring
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with tight nursing follow-up (Experimental): Compared as usual, Patient with tight nursing follow-up will be contacted
  Interventions: Other: tight nursing follow-up
- Patient without tight nursing follow-up (No Intervention): Compared as usual, Patient without tight nursing follow-up will not have interventions

INTERVENTIONS:
Other: tight nursing follow-up — In addition to the usual follow-up by their rheumatologist tight nursing follow-up patients will benefit of
  1. a training session to self-assess their RA: Self-assessment of the number of painful and swollen joints, of pain and disease activity (global assessment by the patient) (self-DAS). During this session, a scheduled dosage of ESR and CRP levels will be given to the patient.
  2. A monthly call by a nurse who inquires about the results of the patient's self-assessment. As soon as she suspects a relapse of RA, she plans a consultation to confirm or not the relapse. For this purpose, she calculates the DAS28 taking into account the results of the biological test, the articular count and the disease activity. Clinical relapse is documented by a DAS28-CRP > 2.7
  Arms: Patient with tight nursing follow-up

SUMMARY:
Rheumatoid arthritis (RA) is a progressive disease that affects mainly small and medium joints and, in the absence of appropriate background therapy, leads to progressive joint destruction, functional, psychological, social and occupational repercussions.

Several biomedicine treat this pathology, including rituximab (RTX). It is recommended to evaluate the therapeutic response to RTX and re-administer it from the 24th week when the goal of remission has not been achieved. However, the optimal modality for reprocessing remains to be determined.

To this end, different approaches have been explored, such as lymphocyte typing or ultrasound monitoring. The pace of these examinations, however, remains wide and their cost is not negligible. This is why we propose here to explore the track of a tight follow-up nurse DAS28.

The hypothesis is that a tight nursing follow-up can detect the symptomatic recovery earlier than the current medical follow-up.

The hypothesis is that a tight nursing follow-up can detect the symptomatic recovery earlier than the current medical follow-up

ELIGIBILITY:
Inclusion Criteria:

* Male or female (age 18 or older)
* Rheumatoid arthritis fulfilling the ACR/EULAR 2010 criteria
* Patient to whom the rheumatologist prescribed a treatment with rituximab or who received a treatment with rituximab in the last 6 months
* Patients with active rheumatoid arthritis prior to treatment with rituximab (DAS 28 CRP>2.7)
* Patient with a DAS 28 CRP of less than 2.7 at 6 months from the last administration of rituximab

Exclusion Criteria:

* Patient not responding to the last treatment with rituximab (DAS28 CRP> 2.7 at 6 months)
* Patient under the age of 18
* Patient with chronic pain due to another pathology than rheumatoid arthritis, which may interfere with the assessment
* Patient with a contraindication to treatment with rituximab
* Woman of childbearing age not taking effective contraception
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Difference from baseline of disease activity specific score | Every 3 months during 2 years
  The disease activity specific score is DAS28-CRP

SECONDARY OUTCOMES:
Difference from baseline in quality of life | Every 3 months during 2 years
  quality of life will be based on HAQ and SF36 questionnaire
Number of cumulative dose of corticosteroids drugs received | Every 3 months during 2 years
Number of cumulative dose of non-steroidal anti-inflammatory drugs received | Every 3 months during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VITTECOQ, Pr, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No